CLINICAL TRIAL: NCT01949961
Title: Randomised Trial of Contrast-enhanced Sonothrombolysis in Acute Ischaemic Stroke
Brief Title: The Norwegian Sonothrombolysis in Acute Stroke Study Part 2
Acronym: NOR-SASS 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding for researchers
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Sykehuset Telemark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REK 2011/2448; 2012-000323-41 (EudraCT Number)
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2018-08

CONDITIONS: Ischemic Stroke
Keywords: intervention; sonothrombolysis; Ultrasound treatment
MeSH Terms: conditions — Ischemic Stroke | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: PROBE: Prospective randomized open-label blinded-endpoint
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound (Active Comparator): Patients eligible (NOR-SASS A/B) and ineligible (NOR-SASS C) for intravenous thrombolysis all receive intravenous ultrasound contrast (microbubbles). The groups are separately randomised to 2 megahertz (MHz) transcranial ultrasound treatment for one hour.
  Interventions: Other: Ultrasound
- Sham ultrasound (Placebo Comparator): Patients eligible (NOR-SASS A/B) and ineligible (NOR-SASS C) for intravenous thrombolysis all receive intravenous ultrasound contrast (microbubbles). The two groups are separately randomised to sham ultrasound treatment for one hour.
  Interventions: Other: Sham ultrasound

INTERVENTIONS:
Other: Ultrasound — SonoVue solution 10 ml (2 vials / 80 µl microbubbles) is given as an infusion of 0,3 ml/min for ~30 minutes, using a Bracco infusion pump.
  Arms: Ultrasound
Other: Sham ultrasound — Mounting the ultrasound headframe but connecting this to a non-operative channel
  Arms: Sham ultrasound

SUMMARY:
BACKGROUND: Thrombolytic drugs may dissolve blood vessel clots in acute ischemic stroke. The overall benefit of intravenous thrombolysis is substantial, but up to 2/3 of patients with large clots may not achieve re-opening of the vessel and up to 40% of the patients may remain severely disabled or die. Ultrasound accelerates clot break-up (lysis) when combined with thrombolysis (sonothrombolysis) and increases the likelihood of functional independence at 3 months. Adding intravenous ultrasound contrast (gaseous microspheres) further enhances the thrombolytic effect (contrast enhanced sonothrombolysis = CEST). Contrast enhanced ultrasound may also accelerate clot break-up in the absence of thrombolytic drugs (contrast enhanced sonolysis = CES).

HYPOTHESIS: Contrast enhanced ultrasound treatment administered within 4 1/2 hours after symptom onset may be given safely to patients with acute ischemic stroke, both to those receiving intravenous thrombolysis and those not receiving intravenous thrombolysis, and will improve clinical outcome.

AIMS: To compare efficacy and safety of contrast enhanced ultrasound treatment vs. no ultrasound treatment in patients with acute ischemic stroke receiving or not receiving intravenous thrombolysis.

STUDY ENDPOINTS: The primary endpoints are 1) neurological improvement at 24 hours (proof of concept) and 2) excellent clinical outcome at 3 months (effect). Secondary endpoints are bleeding complications (safety), brain damage (infarct size/location) and early clinical improvement (effect).

DETAILED DESCRIPTION:
NOR-SASS aims at testing contrast enhanced sonothrombolysis in all patients with acute ischemic stroke. Patients eligible for thrombolysis (randomized tenecteplase or alteplase) are included in the NOR-SASS A sub-study, patients receiving standard (non-trial) thrombolysis with alteplase are included in the NOR-SASS B sub-study, and patients not eligible for thrombolysis are included in the NOR-SASS C sub-study.

DESIGN: NOR-SASS is a PROBE (prospective randomised, open-label, blinded endpoint) trial, designed to establish the superiority of contrast-enhanced ultrasound treatment given within 4½ hours after stroke onset in consecutively admitted patients with acute ischaemic stroke, as compared with 1) standard iv thrombolysis with tenecteplase (TNK) or alteplase (tPA) in patients eligible for thrombolytic treatment, and 2) no specific treatment in patients not eligible for thrombolytic treatment.

HYPOTHESIS: 1.) In patients eligible for intravenous thrombolysis, contrast enhanced sonothrombolysis (CEST) has superior effect as compared with standard intravenous thrombolysis and may be given safely. 2.) In patients not eligible for thrombolysis, contrast enhanced sonolysis (CES) has superior effect as compared with no specific treatment and may be given safely.

RANDOMISATION: In NOR-SASS-A (two step randomisation), 1st randomisation is 1:1 to either tenecteplase (TNK) or alteplase (tPA); 2nd randomisation is 1:1 to either CEST or no CEST. In NOR-SASS-B, randomisation is 1:1 to either CEST or no CEST. In NOR-SASS-C, randomisation is 1:1 to either CES or no CES.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke in the anterior circulation
* Treatment within 4.5 hours after stroke onset
* Informed consent

Exclusion Criteria:

* Patients with premorbid modified Rankin Scale (mRS) score ≥3;
* Patients for whom a complete NIH Stroke Score cannot be obtained;
* Hemiplegic migraine with no arterial occlusion on baseline CT;
* Seizure at stroke onset and no visible occlusion on baseline CT;
* Intracranial haemorrhage on baseline CT;
* Clinical subarachnoid haemorrhage even if baseline CT is normal;
* Large areas of hypodense ischaemic changes on baseline CT;
* Patients with primary endovascular treatment;
* Female, pregnant or breast feeding; pericarditis; sepsis; any other serious medical illness likely to interact with treatment; confounding pre-existent neurological or psychiatric disease; unlikely to complete follow-up; any investigational drug <14 days;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical: Functional handicap | 90 days
  Sliding dichotomy/responder analysis: Excellent outcome is defined as modified Rankin Scale (mRS) 0 with baseline National Institutes of Health Stroke Scale (NIHSS), as mRS 0-1 with baseline NIHSS 8-14, as mRS 0-2 with baseline NIHSS ≥15
Proof of concept: Early neurological improvement | 22-36 hours
  NIHSS=0 or reduction of ≥4 NIHSS points compared with baseline

SECONDARY OUTCOMES:
Symptomatic intracerebral hemorrhage | 24-36 hours
  Local or remote parenchymal haemorrhage type 2 on the 22-36 h post-treatment imaging scan, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline or from the lowest NIHSS value between baseline and 24 h, or leading to death (SITS-MOST criteria).
Hemorrhagic transformation | 24-36 hours
  Any hemorrhagic changes (infarct or parenchymal hematoma)
Short term functional outcome | 7 days
  Sliding dichotomy/responder analysis: Excellent outcome is defined as mRS 0 with baseline NIHSS ≤7, as mRS 0-1 with baseline NIHSS 8-14, as mRS 0-2 with baseline NIHSS ≥15
Brain infarct size and location | 22-36 hours
  MRI infarct volume and ASPECTS score

CONTACTS AND LOCATIONS:
Overall Officials: Lars Thomassen, MD PhD Prof., Study Director — Dept. Neurology, Haukeland University Hospital, Bergen, Norway; Christopher E Kvistad, MD, Study Chair — Dept. Neurology, Haukeland University Hospital, Bergen, Norway; Haakon Tobro, MD, Principal Investigator — Dept. Neurology, Sykehuset Telemark, Skien
Locations (1):
- Dept. of Neurology, Telemark Hospital, Skien, Norway

REFERENCES:
- [Background] Nacu A, Kvistad CE, Logallo N, Naess H, Waje-Andreassen U, Aamodt AH, Solhoff R, Lund C, Tobro H, Ronning OM, Salvesen R, Idicula TT, Thomassen L. A pragmatic approach to sonothrombolysis in acute ischaemic stroke: the Norwegian randomised controlled sonothrombolysis in acute stroke study (NOR-SASS). BMC Neurol. 2015 Jul 11;15:110. doi: 10.1186/s12883-015-0359-4. PMID 26162826
- [Background] Nacu A, Kvistad CE, Naess H, Oygarden H, Logallo N, Assmus J, Waje-Andreassen U, Kurz KD, Neckelmann G, Thomassen L. NOR-SASS (Norwegian Sonothrombolysis in Acute Stroke Study): Randomized Controlled Contrast-Enhanced Sonothrombolysis in an Unselected Acute Ischemic Stroke Population. Stroke. 2017 Feb;48(2):335-341. doi: 10.1161/STROKEAHA.116.014644. Epub 2016 Dec 15. PMID 27980128